CLINICAL TRIAL: NCT05864703
Title: Evaluation of Instantaneous Changes in EEG Activation Patterns Following Application of a Chiropractic Adjustment to the Cervical Spine
Brief Title: Instantaneous EEG Changes Following Chiropractic Adjustment or Sham
Acronym: INS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Reviewing protocol
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: I-0024
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Subluxation
Keywords: Chiropractic; EEG; ECG; sham
MeSH Terms: conditions — Joint Dislocations | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Randomized, sham-controlled trial
Who Masked: Participant
Masking Description: Blind to intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjustment (Experimental): Individuals with a subluxation who receive a true chiropractic adjustment
  Interventions: Procedure: Adjustment
- Sham (Sham Comparator): Individuals with a subluxation who receive a light touch-only sham
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Adjustment — Instrument-assisted, high velocity, low amplitude adjustment
  Arms: Adjustment
Procedure: Sham — Instrument-assisted light touch to neck
  Arms: Sham

SUMMARY:
The project is a randomized, two-arm trial assessing the immediate impact of upper and lower cervical chiropractic adjustments on brain and heart patterns. Thirty individuals (15 per arm) will be recruited from the general population to participate in the study. Qualified participants will undergo a chiropractic physical exam, assessing for cervical subluxations, and a health history review with a Georgia licensed chiropractor. Individuals will be randomized to either an adjustment group or sham group. The adjustment group will receive an upper and lower cervical adjustment with an instrument designed to provide a gentle, targeted adjustment. The sham group will receive a touch sham at similar cervical locations with the same instrument. Both groups will have a 1-hour recording session with an EEG and ECG set-up plus a series of baseline recordings, interventions, and post recordings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18 and 50
* Individuals who can wear an EEG net for 60 minutes Individuals who can sit quietly for at least 20 minutes
* Individuals who can rest on their knees on a massage chair.
* Individuals who have not had a chiropractic adjustment within the last two weeks
* Individuals who have not received any other interventions, such as osteopathic spinal manipulation, physical therapy rehabilitation or manipulation, massage, body movement therapies, or acupuncture within the last two weeks

Exclusion Criteria:

* Individuals who have been diagnosed with a serious mental disorder such as schizophrenia or major depressive disorder that could influence EEG results
* Individuals who do not feel they can sit quietly with limited movement for roughly 20 minutes
* Individuals who cannot rest on their knees on a massage chair.
* Individuals who are on psychotropic medications (e.g. Benzodiazepine medications) that influence EEG readings (Benzodiazepine medications include but are not limited to: alprazolam, chlordiazepoxide, clobazam, clonazepam, clorazepate, diazepam, estazolam, flurazepam, lorazepam, midazolam, oxazepam, temazepam, triazolam, etc.)
* Individuals with any injury or surgery to the skull in the last 6 months, or a history of trauma to the head such as a concussion or stroke
* Individuals who are currently pregnant
* Individuals with a current litigation related to a physical, health-related injury Individuals with untreated diagnosed osteoporosis or articular instability, such as atlanto-axial instability
* Individuals who may require x-rays. Since a single session of chiropractic care is being performed, if at any point the attending chiropractor has any concerns about the ability of the participant to tolerate care or require x-rays, the chiropractor will have the authority to remove the participant from the study.
* Individuals who do not present with a subluxation in the upper cervical region (C1/C2) and in the lower cervical region (C3-C7). The attending chiropractor will determine the presence of the two subluxations during the chiropractic physical exam.
* Individuals with a known heart condition that results in an aberrant ECG recording

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-29 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
EEG resting state effective connectivity | 0 minutes
  Baseline EEG recording for the first intervention or sham procedure. A 64-channel hydronet will be on the head to capture EEG.
EEG resting state effective connectivity | 8 minutes
  EEG recording immediately after the first intervention or sham procedure. A 64-channel hydronet will be on the head to capture EEG.
EEG resting state effective connectivity | 15 minutes
  Baseline EEG recording for the second intervention or sham procedure. A 64-channel hydronet will be on the head to capture EEG.
EEG resting state effective connectivity | 23 minutes
  EEG recording immediately after the second intervention or sham procedure. A 64-channel hydronet will be on the head to capture EEG.

SECONDARY OUTCOMES:
ECG R-R interval | 0 minutes
  Baseline recording for the first intervention or sham procedure. Three leads will on the torso to capture a Lead II ECG.
ECG R-R interval | 8 minutes
  ECG recording immediately after the first intervention or sham procedure. Three leads will on the torso to capture a Lead II ECG.
ECG R-R interval | 15 minutes
  Baseline ECG recording for the second intervention or sham procedure. Three leads will on the torso to capture a Lead II ECG.
ECG R-R interval | 23 minutes
  ECG recording immediately after the second intervention or sham procedure. Three leads will on the torso to capture a Lead II ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, DC, PhD, Study Director — Life University
Locations (1):
- Dr. Sid E. Williams Center for Chiropractic Research, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No